CLINICAL TRIAL: NCT01196195
Title: KONCERT A Kaletra ONCE Daily Randomised Trial of the Pharmacokinetics, Safety and Efficacy of Twice-daily Versus Once-daily Lopinavir/Ritonavir Tablets Dosed by Weight as Part of Combination Antiretroviral Therapy in Human Immunodeficiency Virus-1 (HIV-1) Infected Children (PENTA 18)
Acronym: KONCERT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: Medical Research Council (Other Government); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KONCERT protocol, version 1.6; 2009-013648-35 (EudraCT Number)
Record Dates: First submitted 2010-08-16; First posted 2010-09-08 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Antiretroviral Therapy in HIV-1 Infected Children
Keywords: antiretroviral therapy; child; HIV-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QD kaletra (Experimental): Once daily kaletra
  Interventions: Drug: Kaletra dosed once daily
- BID kaletra (Active Comparator): twice daily dose of kaletra
  Interventions: Drug: kaletra dosed twice daily

INTERVENTIONS:
Drug: Kaletra dosed once daily — Lopinavir/Ritonavir tablets. Dose = 200/50mg or 100/25mg. Frequency = once daily.
  Arms: QD kaletra
Drug: kaletra dosed twice daily — Lopinavir/Ritonavir tablets. Dose = 200/50mg or 100/25mg. Frequency = twice daily.
  Arms: BID kaletra

SUMMARY:
The trial will evaluate the pharmacokinetics, safety, efficacy and acceptability of twice- and once-daily dosing of lopinavir/ritonavir tablets (Kaletra) dosed by weight in HIV-1 infected children who are currently taking lopinavir/ritonavir as part of their combination antiretroviral therapy and who are currently achieving virological suppression (<50 copies/ml). Specifically:

* To confirm weight-based dosing recommendations by evaluating the pharmacokinetics of twice-daily lopinavir/ritonavir half strength formulation tablets dosed on body weight and comparing to historical adult and paediatric data of pharmacokinetics of lopinavir/ritonavir soft gel capsules and oral solution respectively (1, 2).
* To compare the pharmacokinetics of twice-daily lopinavir/ritonavir tablets with once-daily dosing in the same children.
* To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression at 48 weeks. Adherence and acceptability will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* aged <18 years (up to 18th birthday) with confirmed HIV-1 infection
* weight ≥15 kg
* able to swallow tablets
* stable (i.e. CD4 not declining) on a combination antiretroviral regimen that has included lopinavir/ritonavir for at least 24 weeks
* taking lopinavir/ritonavir dosed twice-daily and be willing at the screening visit to change to tablet formulation (if not currently taking tablets) and to change the lopinavir/ritonavir dose to follow the recommended FDA dosing plan based on body weight bands as necessary (see 7.2.2); if participating in the PK study*, be willing at the screening visit to change to lopinavir/ritonavir half strength formulation tablets (100/25mg) only, dosed twice-daily and change the lopinavir/ritonavir dose to follow the recommended FDA dosing plan based on body weight bands as necessary (see 7.2.1)
* viral suppression (HIV-1 RNA <50 copies/ml) for at least the prior 24 weeks (minimum of 2 measurements).
* children and caregivers willing to participate in the PK study if they are among a minimum of the first 16 children enrolled in each body weight band in the trial, including a second PK assessment if randomised to switch to once-daily lopinavir/ritonavir.
* parents/carers and children, where applicable, give informed written consent

Exclusion Criteria:

* children on an antiretroviral regimen that includes a non-nucleoside reverse transcriptase inhibitor (NNRTI), fosamprenavir or nelfinavir
* children who have previously failed virologically on a protease inhibitor (PI) containing regimen (where virological failure is defined as two successive HIV-1 RNA results>1000 copies/ml (confirmed) more than 24 weeks after starting highly active antiretroviral therapy (HAART), i.e changes for toxicity are not counted as failure)
* acute illness
* abnormal renal or liver function (grade 3 or above)
* receiving concomitant therapy except for prophylaxis; Some treatments may be allowed, but must first be discussed with a trial medical expert
* pregnancy or risk of pregnancy in females of child bearing potential

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 173 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed). | week 48
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 Ribonucleic acid (RNA) ≥50 copies/ml (confirmed).
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed). | Week 36
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed).
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed). | week 24
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed).
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed). | week 12
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed).
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed). | week 8
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed).
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed). | week 4
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA ≥50 copies/ml (confirmed).
To compare the pharmacokinetics of twice-daily lopinavir/ritonavir tablets with once-daily dosing in the same children | week 4
  Area under the curve (AUC), minimum observed plasma concentration (Cmin) and maximum observed plasma concentration (Cmax) values of lopinavir after once-daily and twice-daily dosing (in the same children)

SECONDARY OUTCOMES:
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA <400/<50 copies/ml. | week 24
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA <400/<50 copies/ml.
To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA <400/<50 copies/ml. | week 48
  To evaluate whether once-daily dosing of lopinavir/ritonavir is comparable to twice-daily dosing in terms of virological suppression. This is measured by HIV-1 RNA <400/<50 copies/ml.
Acceptability and adherence to once-daily versus twice-daily dosing of lopinavir/ritonavir tablets | week 48
  Acceptability and adherence to once-daily versus twice-daily dosing of lopinavir/ritonavir tablets, assessed by patient/carer completed questionnaires

CONTACTS AND LOCATIONS:
Locations (17):
- Germany (4):
  - Charite University Hospital Berlin, Berlin
  - Department of Pediatric Oncology Hematology and Immunology KA02, Düsseldorf
  - J W Goethe University, Frankfurt
  - Immundefekt-Ambulanz, Dr. von Haunersches Kinderspital, Munich
- Our Lady's Children's Hospital, Dublin, Ireland
- Netherlands (2):
  - Emma Childrens Hospital, Amsterdam
  - UMC St. Radboud, Nijmegen
- Thailand (2):
  - Program for HIV Prevention and Treatment (PHPT)/IRD 174, Changklan, Muang, Chiang Mai
  - HIV-NAT Thai Red Cross AIDS Research Centre, Bangkok
- United Kingdom (8):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospital Bristol, Bristol
  - Evelina Children's Hospital, London
  - Great Ormond Street Hospital, London
  - King's College Hospital, London
  - St. Mary's Hospital, London
  - Nottingham City Hospital Campus, Nottingham
  - John Radcliffe Hospital, Oxford

REFERENCES:
- See also: Related Info — http://www.pentatrials.org/